CLINICAL TRIAL: NCT03346785
Title: The Effect of Social Media Use on Eating Behaviours
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yale-NUS College (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YNC-CPST-02
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Food Photography; Non-Food Photography; No Phone Use
Keywords: External eating; Technology; Photography; Social media

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Food Photography (Experimental): Participants will engage in food photography on their smart phones while eating
  Interventions: Behavioral: Food Photography
- Non-Food Photography (Experimental): Participants will engage in non-food photography on their smart phones while eating
  Interventions: Behavioral: Non-Food Photography
- No Phone Use (Experimental): Participants will not use their smart phones while eating
  Interventions: Behavioral: No Phone Use

INTERVENTIONS:
Behavioral: Food Photography — Participants will engage in food photography on their smart phones while eating
  Arms: Food Photography
Behavioral: Non-Food Photography — Participants will engage in non-food photography on their smart phones while eating
  Arms: Non-Food Photography
Behavioral: No Phone Use — Participants will not use their smart phones while eating
  Arms: No Phone Use

SUMMARY:
This project aims to explore how social media use, in particular food photography, influences eating behaviours. It will be approached through three methods - a correlational experience sampling method, an experimental experience sampling method, and an experimental laboratory method. This registration describes the experimental experience sampling method.

DETAILED DESCRIPTION:
This project aims to explore how social media use, in particular food photography, influences eating behaviours.

The research question will be approached using a combination of methods. The first is the experience sampling method, where data is gathered from participants as they are going about their day-to-day lives. This method comprises two sub-sections - a correlational study, and an experimental study. This registration describes the experimental experience sampling method.

The study will experimentally control participants' engagement in the act of food photography, and measure their eating behaviours. Participants will be recruited via online platforms and participate in the study for one week. At the beginning of the week, they will be required to fill in some online questionnaires (e.g. demographic information). For the rest of the week, they will be prompted at specific time points in the day via smartphone to engage in food photography/ non-food photography/ no phone use, and then answer some questions about their eating behaviours.

The expected outcome of the project is to collectively evaluate the data from the various methods to conclude how social media use, and in particular the act of food photography, influences the various aspects of eating behaviours.

ELIGIBILITY:
Exclusion Criteria:

* Symptoms / history of any medical or psychiatric conditions
* Allergies to food products
* History of eating disorders
* Excessive exercise (≥ 5 times a week of self-reported exercise)
* Currently on a special diet or deliberating restricting caloric intake
* Currently on a weight loss program

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-04-06 (Estimated); Study Completion 2018-04-06 (Estimated)

PRIMARY OUTCOMES:
Enjoyment of food consumed | 15 minutes
  Self-reported rating between 1-7, where 1 is not at all and 7 is very much

SECONDARY OUTCOMES:
Amount of food consumed | 15 minutes
  Self-reported rating between 1-7, where 1 is less than normal and 7 is more than normal

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

REFERENCES:
- [Derived] Yong JYY, Tong EMW, Liu JCJ. Meal-time Smartphone Use in an Obesogenic Environment: Two Longitudinal Observational Studies. JMIR Mhealth Uhealth. 2021 May 6;9(5):e22929. doi: 10.2196/22929. PMID 33955842